CLINICAL TRIAL: NCT01788995
Title: A Non-interventional Trial With Avastin as Front-line Treatment for Ovarian Cancer
Brief Title: BOVARI: A Non-Interventional Study of Avastin (Bevacizumab) as Front-Line Treatment in Patients With Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28355
Record Dates: First submitted 2013-02-08; First posted 2013-02-11 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Ovarian Cancer, Peritoneal Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms; Peritoneal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This non-interventional study will evaluate the routine use and the safety and efficacy of Avastin (bevacizumab) as first-line treatment in patients with advanced ovarian cancer (epithelial ovarian cancer, fallopian tube carcinoma, primary peritoneal carcinoma). Newly diagnosed patients who are initiated on carboplatin/paclitaxel chemotherapy in combination with Avastin will be followed for up to 15 months of treatment and 12 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Patients with newly diagnosed advanced epithelial ovarian cancer (EOC), fallopian tube carcinoma (FTC) or primary peritoneal carcinomas (PPC) with indication for first-line carboplatin/paclitaxel chemotherapy in combination with Avastin

Exclusion Criteria:

* Contraindications for Avastin according to the Summary of Product Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed ovarian cancer (epithelial ovarian cancer, fallopian tube carcinoma or primary peritoneal carcinomas) with indication for carboplatin/paclitaxel chemotherapy in combination with Avastin
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2012-10-15 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
Clinical/demographic patient characteristics at initiation of treatment | approximately 4 years
Duration of treatment | approximately 4 years
Treatment discontinuations/modifications | approximately 4 years

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | approximately 4 years
Progression-free survival | approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Tiroler Landeskrankenanstalten Ges.M.B.H.; Abt. Für Gynäkologie, Innsbruck, Austria